CLINICAL TRIAL: NCT03029182
Title: Simulated-Altitude as an Adjunct to Optimize Aerobic Exercise in Obese Breast Cancer Survivors With Limited Ambulatory Function: Pilot Randomized Trial
Brief Title: Simulated-altitude to Optimize Aerobic Exercise Among Breast Cancer Survivors With Limited Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F160215001
Record Dates: First submitted 2017-01-12; First posted 2017-01-24 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Breast Cancer
Keywords: Exercise; Cancer; Obesity
MeSH Terms: conditions — Obesity; Breast Neoplasms; Motor Activity; Neoplasms | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking+simulated-altitude (Experimental): 8-week exercise training program that involves 3 supervised, treadmill walking sessions each week with 16% oxygen, which will be administered through an exercise mask.
  Interventions: Other: Walking+simulated-altitude
- Walking (control) (Active Comparator): 8-week exercise training program that involves 3 supervised, treadmill walking session each week.
  Interventions: Behavioral: Walking (control)

INTERVENTIONS:
Other: Walking+simulated-altitude — Participants will walk on a treadmill for up to 50 minutes at a 16% oxygen level (administered via exercise mask), which is similar in altitude to Flagstaff, AZ. The progression of exercise training will be based on a varying percents of heart rate reserve.
  Arms: Walking+simulated-altitude
Behavioral: Walking (control) — Participants will walk on a treadmill for up to 50 minutes.The progression of exercise training will be based on a varying percents of heart rate reserve.
  Arms: Walking (control)

SUMMARY:
The study will evaluate the utility of hypoxic exercise training to improve cardiovascular and metabolic health among obese breast cancer survivors. While participants exercise, a lower fraction of inspired oxygen will be used to simulate a higher altitude. This approach removes the mechanical strain needed to sustain moderate-to-vigorous exercise intensity which is believed to support exercise tolerance. Participants are randomized to either the treatment (walking+simulated-altitude) or control (walking under normoxic conditions).

DETAILED DESCRIPTION:
Cancer survivors have a two-fold greater risk of having one or more functional limitations compared to those without a history of cancer. Though exercise interventions in breast cancer survivors exist, a large portion of women (61%) exhibit some form of lower-body dysfunction that severely restricts participation in physical activity and exercise. Both physical and emotional well-being are negatively affected by the combination of increased adiposity, orthopedic problems and muscle weakness, thus reinforcing a cycle of physical inactivity.

For these reasons, obese breast cancer survivors with walking limitations are faced with a barrier that greatly increases the difficulty of meeting prescribed exercise guidelines (≥150 weekly minutes of moderate-to-vigorous intensity exercise). Though previous investigations have demonstrated the safety and benefits of exercise+simulated altitude to improve body fat, physical endurance and insulin sensitivity, results have been limited to non-cancer participants only. Given the comorbidities common to breast cancer survivors, specifically, heart disease risk, lower body joint problems, low aerobic capacity, and fatigue, further research is needed.

ELIGIBILITY:
Inclusion Criteria:

1. Physician's medical clearance for participation
2. English-speaking women
3. 18-70 years of age with a history of Stage 0-III breast cancer
4. Preferred walking speed of less than 2.9 mph as measured by a timed 10 meter walk test (to be performed on-site after consent during preliminary screening) "OR" the inability to complete a 6-minute walk without stopping (to be performed on-site after consent during preliminary screening)
5. Body mass index between 30-45 kg/m2
6. ≥1 year post-treatment and not currently receiving or planning to receive chemo/radiation therapies
7. Not participating in a structured exercise routine
8. In the previous 6 months, not engaging in (on average) ≥60 minutes of moderate or ≥30 minutes of vigorous physical activity per week.

Exclusion Criteria:

1. Males
2. Dementia
3. Medical, psychological, and/or social characteristics that may interfere with the ability to fully participate in the proposed study activities/assessments (e.g., psychosis, schizophrenia)
4. Contraindication to participate in regular exercise training
5. Unwilling to complete prescribed exercise
6. Inability to walk
7. Pregnant
8. Resting oxygen saturation via pulse oximetry below 90%
9. Using home oxygen therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of an 8 week exercise intervention comparing walking+simulated-altitude to walking (control) based on retention. | baseline to 8 weeks
  number of participants completing the 8 week session
Determine the feasibility of an 8 week exercise intervention comparing walking+simulated-altitude to walking (control) based on adherence to exercise compliance. | baseline to 8 weeks
  mean compliance among all participantswith exercise prescription
Determine the feasibility of an 8 week exercise intervention comparing walking+simulated-altitude to walking (control) based on number of adverse events. | baseline to 8 weeks
  Number of adverse events in each group

SECONDARY OUTCOMES:
The effect sizes for walking+simulated-altitude and walking (control) as measured by a 6 minute walk. | baseline to 8 weeks
  6 minute walk test, a valid and reliable tool in cancer survivors will be used to evaluate cardiovascular health and mobility. Total distance (in meters) covered over the duration of 6 minutes will be recorded.
The effect sizes for walking+simulated-altitude and walking (control) as measured by the cardiorespiratory fitness. | baseline to 8 weeks
  Cardiorespiratory fitness, will be measured by indirect calorimetry during a graded walking test on a treadmill to estimate peak aerobic capacity.
The effect sizes for walking+simulated-altitude and walking (control) as measured by arterial elasticity. | baseline to 8 weeks
  Arterial elasticity, will be measured by local pulse contour analyses (HDI/Pulse Wave), A non-invasive procedure based on a modified Windkessel model which permits the evaluation of vascular health.
The effect sizes for walking+simulated-altitude and walking (control) as measured by resting heart rate variability. | baseline to 8 weeks
  Heart rate variability, will be determined by R-to-R interval variations in heart rate, used to index sympatho-vagal balance.
The effect sizes for walking+simulated-altitude and walking (control) as measured by the fasting glucose. | baseline to 8 weeks
  Typically, a "normal" blood sugar level is identified by experts as anything less than 100 mg/dL after a period of fasting.
The effect sizes for walking+simulated-altitude and walking (control) as measured by C-reactive protein (mg/L) serum assays. | baseline to 8 weeks
  Serum assays, will be measured following an overnight to evaluate metabolic and cardiovascular health. Standards practices will be implemented.
The effect sizes for walking+simulated-altitude and walking (control) as measured by tumor-necrosis factor-alpha (pg/mL) assays. | baseline to 8 weeks
  Serum assays, will be measured following an overnight to evaluate metabolic and cardiovascular health. Standards practices will be implemented.
The effect sizes for walking+simulated-altitude and walking (control) as measured by interleukin-6 (pg/mL) serum assays. | baseline to 8 weeks
  Serum assays, will be measured following an overnight to evaluate metabolic and cardiovascular health. Standards practices will be implemented.
The effect sizes for walking+simulated-altitude and walking (control) as measured by interleukin-10 (pg/mL) serum assays. | baseline to 8 weeks
  Serum assays, will be measured following an overnight to evaluate metabolic and cardiovascular health. Standards practices will be implemented.
The effect sizes for walking+simulated-altitude and walking (control) as measured by body composition (% body fat). | baseline to 8 weeks
  Body composition, will be measured by dual-energy X-ray absorptiometry during which participants will be scanned while lying supine in light clothing with their arms at their sides.
The effect sizes for walking+simulated-altitude and walking (control) as measured by free-living physical activity. | baseline to 8 weeks
  Free-living physical activity, will be measured by a triaxial accelerometer (e.g., Actigraph GT3X). Participants will wear the accelerometer on the hip of their non-dominant side during waking periods and around the wrist when sleeping according to a previously published protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States